CLINICAL TRIAL: NCT06423781
Title: A Phase 2, Multicenter, Open-Label Extension Study to Assess the Long-Term Safety and Tolerability of BHV-7000 in Treatment of Major Depressive Disorder (MDD)
Brief Title: Long-term Safety Study of BHV-7000 in Participants With Major Depressive Disorder (MDD)
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHV7000-203
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
Keywords: depression; major depression; antidepressant; major depressive disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BHV-7000 (Experimental)
  Interventions: Drug: BHV-7000

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 75 mg taken once daily

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of BHV-7000, in participants with Major Depressive Disorder (MDD).

ELIGIBILITY:
Key Inclusion Criteria:

1. Eligible subjects should have successfully completed the Treatment/Randomization Phase of parent studies.
2. WOCBP must have a negative urine pregnancy test at Baseline Visit.
3. WOCBP must not be breastfeeding or lactating at Baseline Visit or at any point during the study.

Key Exclusion Criteria:

1. Any medical condition, based on the judgement of the Investigator, that would confound the ability to adequately assess safety and efficacy outcome measures.
2. Participant non-compliance with study procedures, study drug or visit attendance in the parent study that the Investigator deems as clinically significant or unacceptable risk potential for this study.
3. Investigator deems participant at imminent risk of danger to others.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and AEs judged to be related to study medication | Up to 104 weeks
  Safety and tolerability of BHV-7000 as assessed by frequency of unique subjects with SAEs; AEs leading to discontinuation; AEs judged to be related to study medication
Number of Participants With Clinically Significant Laboratory Abnormalities | Up to 104 weeks
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 or 4 laboratory abnormalities.
Number of Participants With Vital Sign Abnormalities | Up to 104 weeks
Number of Participants With Electrocardiogram (ECG) Abnormalities specific to QTc elevation | Up to 104 weeks

CONTACTS AND LOCATIONS:
Locations (66):
- United States (66):
  - Reverie Mind, LLC, Chandler, Arizona
  - IMA Clinical Research, Phoenix, Arizona
  - Pillar Clinical Research, LLC, Little Rock, Arkansas
  - WIRG, Little Rock, Arkansas
  - WRN, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CIT LA, Bellflower, California
  - IPMG, Chino, California
  - WR-PRI Encino, Encino, California
  - Collaborative Neuroscience Research, LLC (CenExel - CNS), Garden Grove, California
  - CalNeuro Research Group, Los Angeles, California
  - Excell Research, Inc., Oceanside, California
  - NRC Research Institute, Orange, California
  - Anderson Clinical Research, Redlands, California
  - CIT IE, Riverside, California
  - Lumos Clinical Research Center, LLC, San Jose, California
  - Stanford, Stanford, California
  - Cenexel CNS, Torrance, California
  - Pacific Clinical Research Management Group, Upland, California
  - Sunwise Clinical Research, Walnut Creek, California
  - MCB Clinical Research Centers, Colorado Springs, Colorado
  - UConn Health, Farmington, Connecticut
  - Optum Behavioral Care of Connecticut, PC dba Comprehensive Psychiatric Care of Connecticut, Norwich, Connecticut
  - Clinical Neuroscience Solutions, Inc, Jacksonville, Florida
  - Floridian Neuroscience Institute, Miami Lakes, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - K2 Medical Research, Tampa, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Revive Research Institute, Inc., Elgin, Illinois
  - Collective Medical Research, Overland Park, Kansas
  - DelRicht Research, New Orleans, Louisiana
  - Headlands Pharmasite, Baltimore, Maryland
  - CBH Health, Gaithersburg, Maryland
  - Copley Clinical, Boston, Massachusetts
  - Boston Clinical Trials, Boston, Massachusetts
  - Adams Clinical, Watertown, Massachusetts
  - Precise Clinical Research, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - IMA Clinical Research, Las Vegas, Nevada
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Bio Behavioral Health, Toms River, New Jersey
  - SPRI Clinical Trials, LLC, Brooklyn, New York
  - Neurobehavioral Research, Inc, Cedarhurst, New York
  - Bioscience Research LLC, Mount Kisco, New York
  - Berman Clinical, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - The Medical Research Network, LLC, New York, New York
  - RBA, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - Summit Headlands LLC, Portland, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Suburban Research Associates, Media, Pennsylvania
  - Scranton Medical Institute, Moosic, Pennsylvania
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Donald J. Garcia, MD, PA dba Austin Clinical Trial Partners, Austin, Texas
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Relaro Medical Trials, LLC, Dallas, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Aim Trials, Plano, Texas
  - Grayline Research Center, Wichita Falls, Texas
  - Alpine Reseach Organization, Clinton, Utah
  - Northwest Clinical Research Center, Bellevue, Washington